CLINICAL TRIAL: NCT07299942
Title: Beta-glucan Supplementation During Calorie and Carbohydrate-restricted Diet: Impact on Body Weight and Body Fat Loss, Subjective Appetite, and Gastrointestinal Appetite Hormones of Healthy Women With Overweight.
Brief Title: Impact of Beta-glucan Supplementation During Calorie and Carbohydrate-restricted Diet on Body Weight and Body Fat Loss, Appetite, and Gastrointestinal Appetite Hormones.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Dalia Malkova, Dr, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200230098
Record Dates: First submitted 2025-05-01; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-10

CONDITIONS: Overweight and Obese Women
Keywords: overweight, obesity, body weigh loss, beta-glucan, appetite
MeSH Terms: conditions — Overweight; Obesity | interventions — Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-glucan (9g/day) supplementation (Experimental): Beta-glucan (9g/day) combined with consumption of low low-calorie and low-carbohydrate diet for four weeks.
  Interventions: Combination Product: Beta-glucan addition to a restricted calorie of meal replacements and carbohydrate diet.
- Cellulose addition to low calorie and low carbohydrate diet. (Placebo Comparator): Cellulose (9g/day) combined with consumption of low low-calorie and low-carbohydrate diet for four weeks.
  Interventions: Combination Product: Cellulose (Placebo) addition to a restricted calorie of meal replacements and carbohydrate diet.

INTERVENTIONS:
Combination Product: Beta-glucan addition to a restricted calorie of meal replacements and carbohydrate diet. — Female participants will undergo a 4-week intervention, which will involve taking 9g/day of beta-glucan supplement while consuming low-calorie liquid meal replacements (Cambridge Weight Plan, Corby, UK) for breakfast and dinner, each providing 200kcal, and low-carbohydrate lunches.
  Arms: Beta-glucan (9g/day) supplementation
Combination Product: Cellulose (Placebo) addition to a restricted calorie of meal replacements and carbohydrate diet. — Female participants will undergo a 4-week intervention, which will involve taking 9 g/day of cellulose while consuming low-calorie liquid meal replacements (Cambridge Weight Plan, Corby, UK) for breakfast and dinner, each providing 200kcal, and low-carbohydrate lunches.
  Arms: Cellulose addition to low calorie and low carbohydrate diet.

SUMMARY:
This study will investigate whether beta-glucan supplementation, when added to an energy and carbohydrate-restricted diet, facilitates body weight and body fat loss, and leads to less detrimental changes in subjective appetite and gastrointestinal appetite hormones. This will be a double-blind, randomised, controlled trial in which healthy females living with overweight and obesity will be randomly assigned to a beta-glucan or a cellulose (placebo) group (1:1 basis). The randomisation software will be used to generate a randomisation list. This list will be held by a person independent of the research team. During the 4-week intervention, participants will consume an energy and carbohydrate-restricted diet combined with 9 g/day of beta-glucan (beta-glucan group) or 9 g/day of cellulose (Placebo group). During the 4-week intervention, breakfasts and dinners will consist of energy-restricted meal replacements providing 200 kcal/ meal, while lunches will be low-carbohydrate meals providing 35% of habitual energy intake. Before and at the end of the intervention, participants will conduct an experimental trial, with pre- and post-intervention trials being identical. The experimental trials will take place in the metabolic room of the New Lister Building (NLB) of the Glasgow Royal Infirmary. During the experimental trials, body weight and body composition will be measured in the fasted state, and the collection of fasting and postprandial (for the duration of 240 minutes) blood samples will be conducted. For a meal, participants will consume the low-calorie breakfast, which will be a liquid meal replacement (Cambridge Weight Plan, Corby, UK), together with 3 g of beta-glucan. Subjective appetite scores will be measured in the fasted and postprandial states. To achieve total body water and thus body composition (fat mass and fat-free mass) measurements, saliva will be collected before and 3 and 3.5 hours after consumption of D2O (which will be consumed in the fasted state). For the duration of 24 hours before the experimental trial, participants will be asked to avoid coffee and alcohol. Participants will be required to record their food and drink intake for three days before the trial days of each experimental investigation.

DETAILED DESCRIPTION:
This study will investigate whether beta-glucan supplementation, when added to an energy and carbohydrate-restricted diet, facilitates body weight and body fat loss, and leads to less detrimental changes in subjective appetite and gastrointestinal appetite hormones. This will be a double-blind, randomised, controlled trial in which healthy females living with overweight and obesity will be randomly assigned to a beta-glucan or a cellulose (placebo) group (1:1 basis).

Participants Based on power calculations and taking into consideration a drop-out rate of approximately 25%, this study will aim to recruit 60 sedentary females living with overweight or obesity (30 in each group), aged between 18 and 60 years and with a body mass index (BMI) between 25 and 39.9 kg/m².

Study design To confirm the eligibility, study participants will undergo a screening session. The screening visit will involve completion of a health questionnaire, height and body weight, and resting metabolic rate measurements. Eligible participants will be randomised either to the beta-glucan or the placebo group. Randomisation will be performed using Excel software. To ensure that the study was blinded, an independent person labelled the packs of fibre as either 'A' or 'B', indicating the β-glucan or placebo group.

Prior to the 4-week intervention, participants will undergo an experimental trial. This trial will be conducted at the Metabolic Investigation Laboratory, beginning at approximately 9:00 am, following an overnight fast. Height and body weight will be measured using the same procedures employed during the screening session. Participants will then complete a subjective appetite questionnaire. After that, a cannula will be placed into the antecubital vein. After a 10-minute rest period, a fasting blood sample will be collected. Following this, a baseline saliva sample will be obtained, and participants will be asked to consume deuterium oxide (D₂O) mixed with regular drinking water. Immediately after the baseline saliva collection, participants will consumed a standardised low-calorie breakfast (~200 kcal; carbohydrates: 20-25 g, protein: 15-20 g, fat: ~3 g, fibre: ~2 g) which will be a liquid meal replacement (Cambridge Weight Plan, Corby, UK), mixed with either 3 g of β-glucan or 3 g of cellulose as a placebo. During the experimental trials, blood samples and subjective appetite scores will be collected at 30-minute intervals for the duration of 240 minutes, and additional saliva samples will be collected at 3 hours and 3.5 hours post-ingestion of deuterium oxide water. The identical trial will be conducted after the intervention completion.

During the 4-week intervention, participants will consume an energy and carbohydrate-restricted diet combined with 9 g/day of beta-glucan (beta-glucan group) or 9 g/day of cellulose (Placebo group). During the 4-week intervention, breakfasts and dinners will consist of energy-restricted meal replacements providing 200 kcal/ meal, while lunches will be low-carbohydrate meals providing 35% of habitual energy intake.

During the intervention, participants will be provided with the supplements (beta-glucan or placebo) and low-energy liquid meal replacement sachets in two separate batches. This approach is expected to support compliance with the study products. Participants were instructed to consume 9 g/day either a beta-glucan or a placebo supplement with each main meal (breakfast, lunch, and dinner). For breakfast and dinner, the fibre will be mixed with the provided meal replacements. For lunch, participants will be advised to mix supplements with yoghurt, juice, or water based on personal preference. Participants will be contacted by telephone or email once a week to provide dietary review and support. Participants will be encouraged to avoid consuming alcohol or to have a maximum of two units per week.

Outcome Measures Fat-free mass (FFM) and fat mass (FM) will be measured in both pre-intervention and post-intervention experimental trials using a stable isotope dilution method with deuterium oxide (D₂O) as a tracer. The amount of D₂O in the body will be analysed using Fourier Transform Infrared Spectrometry.

This technique has been used for the last 50 years to estimate total body water (TBW), which is used to calculate fat-free mass and teh fat mass.

Subjective appetite scores will be measured using the Visual Analogue Scale (VAS). The scale is 100 mm in length with words anchored to a minimum and a maximum of the ''desire to eat'', ''fullness'', ''hunger'', ''capacity to eat'' and ''satiety'' the point corresponding to their sensations. The response will be calculated by measuring the distance in millimeters from the left-hand anchor to the participant's mark. All scores will be completed manually.

Appetite-Related Hormones. The measurements of plasma concentration of total ghrelin, acylated ghrelin, PYY, GLP-1 will be measured using ELISA kits (Merck, Millipore, Bioscience Division, UK).

Dietary assessment. Food diaries and electronic kitchen scales (Salter Housewares Ltd., Tonbridge, UK) will be given to participants on the screening day, and participants will be instructed on how to use the scales to record 3-day food and beverage intake. Dietary records will be analysed for energy and macronutrient intake using the Nutritics dietary analysis software (Dublin, Ireland). The dietary assessment data were used to characterise participants' habitual dietary patterns.

Statistical Analysis. Mixed ANOVA using the general linear model with group (control and β-glucan) will be used for assessing the effect of time, group, and time*group interaction on body weight, fat mass, fat-free mass, composite appetite scores, and gastrointestinal appetite hormones (total ghrelin, PYY and GLP-1).

ELIGIBILITY:
Inclusion Criteria:

* Healthy females living with overweight or obese (BMI of 25 - 39.9 kg/m2).
* Age between 18 to 60 years.
* Stable body weight for at least 3 months preceding the study.

Exclusion Criteria:

* Smokers
* Irregular menstrual cycle
* Exercising more than 75min a week
* Pregnant or lactating
* Food allergies
* Vegan or vegetarian or follow any diet other than the typical Western diet.
* Taking dietary supplement at the time of the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female by birth.
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Body weight | At the beginning (baseline, week 0 ) and at the end of the 4-week intervention, (post, week 4).
  Body weight will be assessed in the fasted state using bioelectrical impedance analysis (TANITA-TBF-310, Cranela, UK).
Total body water | At the beginning (baseline, week 0 ) and at the end of the 4-week intervention (post, week 4).
  Saliva samples collected before and after 3 hours and 3.30 hours of drinking D2O water during experimental trials, which will be conducted before and after 4 week intervention, will be analysed for total body water using Fourier Transform spectroscopy (FTIR).
Subjective appetite | At the beginning (baseline, week 0 ) and at the end of the 4-week intervention (post, week 4).
  Assessment of fasting and postprandial (over a duration of 240 minutes) appetite via visual analogue scale (100mm) during the experimental trials, conducted before (week 0) and after 4 4-week intervention.

SECONDARY OUTCOMES:
Gastrointestinal appetite hormones | At the beginning (baseline, week 0 ) and at the end of the 4-week intervention (post, week 4).
  Fasting and postprandial (over duration of 240 minutes) blood collection during the experimental trials, conducted before and after 4 week intervention, for the measurements of ghrelin, acylated ghrelin, GLP-1, PYY concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition, College of Medicine, Veterinary and Life Science,, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This study will published in scientific journals when is finished

REFERENCES:
- See also: Related Info — https://doi.org/10.1017/S0029665124004543